CLINICAL TRIAL: NCT05319262
Title: Metabolic and Cognitive Consequences of Noise-induced Sleep Disturbance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: University of Pennsylvania (Other); University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 234826201
Record Dates: First submitted 2022-03-09; First posted 2022-04-08 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Noise Exposure; Sleep Disturbance; Sleep Hygiene; Metabolic Disturbance; Cognitive Change
Keywords: neurobehavioral performance; white noise; auditory fatigue; polysomnography; metabolomics
MeSH Terms: conditions — Parasomnias; Sleep Hygiene

STUDY DESIGN:
Intervention Model Description: All participants will be exposed to each of the different noise exposure conditions. Each study night is treated as a separate arm of the crossover study. The order of the noise exposure conditions will be be randomly assigned across participants using a Latin square design to avoid first-order carryover effects. Each subject will be exposed to one night of each of the following:
  Quiet night: No noise will be played, serving as a control night to assess individual baseline sleep, metabolic profile, and cognitive performance; Traffic noise night to determine consequences of noise-disrupted sleep; Pink noise night: To determine impact of continuous pink noise on sleep; Traffic + pink noise night: simultaneous traffic and pink noise at the same sound pressure levels as in the traffic-only and pink noise-only nights, to determine sleep-protecting effects of pink noise in the face of traffic noise.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be aware that in any given study night they can be exposed to traffic noise and/or pink noise. They will not be informed what noise condition will occur in any given night, but they can become unblinded to the exposure if they are awake, as they will hear the noise.
  Study investigators responsible for analysing cognitive performance variables and physiological sleep data will be be blind to which noise interventions were introduced on which study nights.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Single study night with no noise exposure, to determine normal baseline sleep
- Traffic noise (Experimental): Single study night with traffic noise events, to determine consequences of sleep disturbance by traffic noise
  Interventions: Radiation: Traffic noise
- Pink noise (Experimental): Single study night to measure the effects of a non-pharmacological intervention to promote sleep, pink noise.
  Interventions: Radiation: Pink noise exposure
- Traffic noise + pink noise (Experimental): Single study night with concurrent traffic noise events and continuous pink noise sound exposure. Night is used to determine attenuation of sleep disturbance by traffic noise due to introduction of pink noise.
  Interventions: Radiation: Pink noise exposure; Radiation: Traffic noise

INTERVENTIONS:
Radiation: Pink noise exposure — Continuous pink noise sound exposure at 45 dBA, throughout the whole night
  Arms: Pink noise; Traffic noise + pink noise
Radiation: Traffic noise — 120 traffic noise events (40 each of road, rail and aircraft), introduced at maximum sound pressure levels ranging between 45-65 dB LAS.max.
  Arms: Traffic noise; Traffic noise + pink noise

SUMMARY:
This study will investigate the biological mechanisms linking sleep disruption by noise and the development of disease. In a laboratory sleep study, we will play traffic sounds of different types (road, rail and air) and noise levels during the night. We will also have nights with sound from so-called "white noise machines". These generate a low-level and continuous noise that may improve sleep by "masking" the traffic noises that would otherwise disturb sleep. We will also measure objective sleep quality and quantity, cognitive performance across multiple domains, self-reported sleep and wellbeing outcomes, and blood samples. Blood samples will be analysed to identify metabolic changes in different nights. Identifying biomarkers that are impacted by sleep fragmentation will establish the currently unclear pathways by which chronic noise exposure at night can lead to the development of diseases in the long term, especially cardiometabolic disorders.

DETAILED DESCRIPTION:
The experimental sleep study has the overarching goal of deepening our understanding of experimentally-induced disruption of sleep and changes in metabolic and cognitive function, and to determine the efficacy of a potential non-pharmacological intervention to promote sleep. To this end, the study will address the following independent aims:

Aim 1: Determine associations between novel physiologic markers of sleep and metabolic and cognitive function. We will measure the sleep of healthy volunteers using novel and classical indictors of sleep architecture. Each morning we will obtain blood samples for metabolomics analysis and administer a neurocognitive test battery.

Aim 2: Determine the biological and neurobehavioral consequences of noise-disrupted sleep. We will compare effects on sleep, metabolomics and cognitive function between quiet nights and nights with traffic noise.

Aim 3: Evaluate the effects of continuous pink noise throughout the night. Sub-aim 1: To determine if continuous noise (pink noise) per se improves or disturbs sleep, we will investigate changes in novel and classical indictors of sleep architecture and disturbance induced by pink noise relative to quiet baseline nights. Sub-aim 2: To determine if pink noise reduces sleep disturbance by traffic noise, we will investigate changes in sleep fragmentation and continuity, and cortical and autonomic arousal, from nights with both traffic noise and pink noise compared to nights with traffic noise only.

The study will be conducted at in the University of Gothenburg sound environment laboratory (SEL). The SEL is a high fidelity research laboratory equipped to simulate a typical apartment, including three individually light-, sound- and vibration-isolated private bedrooms. Ceiling mounted speakers in each room allow us to create a realistic acoustic environment by transmitting sound exposures from the control room to each bedroom individually.

This study has a prospective within-subjects cross-over design. Participants (N=12) will each spend five consecutive nights in the SEL with a sleep opportunity between 23:00-07:00. Daytime sleep will be prohibited, confirmed with measures of daytime activity via wrist actigraphy monitors worn continuously throughout the study. Three subjects will take part concurrently, in separate bedrooms. The first night is a habituation period to the study protocol and for familiarisation with the test procedures. Study nights 2-5 are the experimental nights and will be randomly assigned across participants using a Latin square design to avoid first-order carryover effects. Each subject will be exposed to one night of each of the following:

Quiet night: No noise will be played, serving as a control night to assess individual baseline sleep, metabolic profile, and cognitive performance; Traffic noise night to determine consequences of noise-disrupted sleep; Pink noise night: To determine impact of continuous pink noise on sleep; Traffic + pink noise night: simultaneous traffic and pink noise at the same sound pressure levels as in the traffic-only and pink noise-only nights, to determine sleep-protecting effects of pink noise in the face of traffic noise.

Each night we will record physiologic sleep with polysomnography (PSG) and cardiac activity with electrocardiography (ECG). Each study morning, subjects will provide a 2ml blood sample, complete cognitive testing and answer questionnaires and will depart the SEL to follow their normal daytime routine. They will return to the SEL at 20:00 each evening to prepare for sleep measurements. Caffeine will be prohibited after 15:00 and alcohol will be prohibited at all times. Because sound-induced auditory fatigue may be affected by noise exposure during participant's normal routines,60 they will wear a noise dosimeter during the week of the study to record their daytime noise exposure. Because extreme and/or variable dietary behaviour can affect the metabolome/lipoprotein profile, participants will be given guidance that they should eat a similar evening meal on each day of the laboratory study, confirmed with a food diary, The actual meal itself can be different for different study participants, because the study has a within-subjects design.

Sleep will be recorded with ambulatory polysomnography (PSG) and cardiac activity with electrocardiography (ECG) and finger pulse photoplethysmogram. Data are recorded offline onto the sleep recorder, and will be downloaded and checked every study morning to ensure data quality. In addition to traditional sleep analysis performed by the research group at the University of Gothenburg, raw PSG data will be used to calculate the Odds Ratio Project, a novel metric of sleep depth and stability.

Each study morning subjects will provide a 2 ml blood sample for plasma metabolomics analysis. To ensure reliable data, blood samples will be taken at the same time every day to mitigate circadian effects, before eating or drinking anything except water, and each sample will be handled in the same way i.e. centrifuged, aliquoted and stored in -80C freezers. Subjects will eat the same food each study evening to mitigate within-subject dietary effects on the blood metabolome.

Each morning, subjects will complete a computerised cognitive test battery taking approximately 20 minutes, that includes 10 tests across a range of cognitive domains (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance). Cognition data will be analysed to determine key measures of cognitive speed and accuracy, adjusting for practice effects and the difficulty of the stimulus set.

Subjects will complete a battery of one-time validated questionnaires to measure their general health (SF-36), chronotype, noise sensitivity, habitual sleep quality, environmental sensitivity, and annoyance and sleep disturbance by noise. Subjects will also answer a questionnaire each study evening and morning, involving questions on sleepiness (Karolinska Sleepiness Scale), auditory fatigue, sleep disturbance by noise, and validated sleep and disturbance questions.

Subjects will wear a noise dosimeter during the week of the study to record their daytime noise exposure (sound pressure level only, no actual sound recordings).

Participants will wear a wrist actigraphy monitor continuously throughout the study period, and also for the week before the study, to confirm habitual sleep-wake times and to measure physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

1) live in or around the city of Gothenburg area (Sweden)

Exclusion Criteria:

1. aged <18 or >30 years;
2. habitual sleep and wake timings more than ±1 hour different from the study sleep times (i.e. habitual sleep time should be 22:00-00:00 and habitual wake time should be 06:00-08:00);
3. BMI>25 kg/m2;
4. regular sleep medication use (prescribed or "over-the-counter");
5. poor hearing acuity (measured during screening via pure tone audiometry);
6. diagnosed with sleep disorders;
7. indications of sleep apnea on the STOP-BANG questionnaire;
8. shift work;
9. smoking, vaping, snus, or other nicotine use;
10. pre-existing use of "white noise machines" as a sleep aid.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-04-24 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Metabolomics and lipids | On each of the five study mornings
  Concentrations of 41 metabolites, including amino acids, amines, alcohols, carboxylic acids, choline, keto acids, sugars, and sulfones. Lipoprotein profile, including concentrations of triglycerides, cholesterol, phospholipids, and apolipoproteins.
Baseline total sleep time | During the Control night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total sleep time during exposure to nocturnal traffic | During the traffic noise night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total sleep time during exposure to pink noise | During the pink noise night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total sleep time during exposure to traffic noise + pink noise | During the Traffic noise + pink noise night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of baseline N1 sleep | During the Control night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of baseline N2 sleep | During the Control night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of baseline N3 sleep | During the Control night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of baseline rapid eye movement (REM) sleep | During the Control night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N1 sleep during exposure to nocturnal traffic | During the traffic noise night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N2 sleep during exposure to nocturnal traffic | During the traffic noise night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N3 sleep during exposure to nocturnal traffic | During the traffic noise night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of rapid eye movement (REM) sleep during exposure to nocturnal traffic | During the traffic noise night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N1 sleep during exposure to pink noise | During the pink noise night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N2 sleep during exposure to pink noise | During the pink noise night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N3 sleep during exposure to pink noise | During the pink noise night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of rapid eye movement (REM) sleep during exposure to pink noise | During the pink noise night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N1 sleep during exposure to traffic noise + pink noise | During the Traffic noise + pink noise night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N2 sleep during exposure to traffic noise + pink noise | During the Traffic noise + pink noise night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N3 sleep during exposure to traffic noise + pink noise | During the Traffic noise + pink noise night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of rapid eye movement (REM) sleep during exposure to traffic noise + pink noise | During the Traffic noise + pink noise night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Baseline wakefulness after sleep onset (WASO) | During the Control night
  Total number of minutes awake during the night after the first appearance of sleep of any stage. Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Wakefulness after sleep onset (WASO) during exposure to nocturnal traffic | During the Traffic noise night
  Total number of minutes awake during the night after the first appearance of sleep of any stage. Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Wakefulness after sleep onset (WASO) during exposure to pink noise | During the Pink noise night
  Total number of minutes awake during the night after the first appearance of sleep of any stage. Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Wakefulness after sleep onset (WASO) during exposure to traffic noise + pink noise | During the Traffic noise + pink noise night
  Total number of minutes awake during the night after the first appearance of sleep of any stage. Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Baseline number of awakenings | During the Control night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Number of awakenings during exposure to nocturnal traffic | During the Traffic noise night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Number of awakenings during exposure to pink noise | During the Pink noise night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Number of awakenings during exposure to traffic noise + pink noise | During the Traffic noise + pink noise night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Baseline sleep onset latency (SOL) | During the Control night
  Defined as the time from lights out to the first epoch of sleep measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep onset latency (SOL) during exposure to nocturnal traffic | During the Traffic noise night
  Defined as the time from lights out to the first epoch of sleep measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep onset latency (SOL) during exposure to pink noise | During the Pink noise night
  Defined as the time from lights out to the first epoch of sleep measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep onset latency (SOL) during exposure to nocturnal traffic and pink noise | During the Traffic noise + Pink noise night
  Defined as the time from lights out to the first epoch of sleep measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Baseline sleep efficiency | During the Control night
  Defined as the percentage of time in bed spent in a non-wake sleep stage, measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep efficiency during exposure to nocturnal traffic | During the Traffic noise night
  Defined as the percentage of time in bed spent in a non-wake sleep stage, measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep efficiency during exposure to pink noise | During the Pink noise night
  Defined as the percentage of time in bed spent in a non-wake sleep stage, measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep efficiency during exposure to nocturnal traffic and pink noise | During the Traffic noise + pink noise night
  Defined as the percentage of time in bed spent in a non-wake sleep stage, measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Baseline sleep depth assessed using the odds ratio product (ORP) | During the Control night
  Average ORP over the full night, from 0 (never occurs during wake) to 2.5 (only occurs during wake). Derived via polysomnography/EEG measurements.
Sleep depth assessed using the odds ratio product (ORP) during exposure to nocturnal traffic | During the Traffic noise night
  Average ORP over the full night, from 0 (never occurs during wake) to 2.5 (only occurs during wake). Derived via polysomnography/EEG measurements.
Sleep depth assessed using the odds ratio product (ORP) during exposure to pink noise | During the Pink noise night
  Average ORP over the full night, from 0 (never occurs during wake) to 2.5 (only occurs during wake). Derived via polysomnography/EEG measurements.
Sleep depth assessed using the odds ratio product (ORP) during exposure to traffic noise and pink noise | During the Traffic noise + pink noise night
  Average ORP over the full night, from 0 (never occurs during wake) to 2.5 (only occurs during wake). Derived via polysomnography/EEG measurements.
Spontaneous maximal change of odds ratio product (ORP) | During the Control night
  Primary measure of acute sleep disruption by noise, calculated as the difference between the ORP in the 30s prior to noise onset and the maximum ORP during traffic noise. Averaged over 120 sham noise events during the night.
Maximal change of odds ratio product (ORP) during exposure to traffic noise events | During the Traffic noise night
  Primary measure of acute sleep disruption by noise, calculated as the difference between the ORP in the 30s prior to noise onset and the maximum ORP during traffic noise. Averaged over all 120 noise events during the night.
Maximal change of odds ratio product (ORP) during exposure to traffic noise events | During the Traffic noise + pink noise night
  Primary measure of acute sleep disruption by noise, calculated as the difference between the ORP in the 30s prior to noise onset and the maximum ORP during traffic noise. Averaged over all 120 noise events during the night.
Spontaneous change of odds ratio product (ORP) during exposure to pink noise | During the Pink noise night
  Primary measure of acute sleep disruption by noise, calculated as the difference between the ORP in the 30s prior to noise onset and the maximum ORP during traffic noise. Averaged over 120 sham noise events during the night.
Baseline morning neurobehavioural speed | In the morning immediately after the Control night
  Average of one key speed indicator from each of 10 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance)
Morning neurobehavioural speed after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Average of one key speed indicator from each of 10 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance)
Morning neurobehavioural speed after exposure to pink noise | In the morning immediately after the Pink noise night
  Average of one key speed indicator from each of 10 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance)
Morning neurobehavioural speed after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Average of one key speed indicator from each of 10 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance)
Baseline morning neurobehavioural accuracy | In the morning immediately after the Control night
  Average of one key accuracy indicator from each of 9 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, psychomotor vigilance)
Morning neurobehavioural accuracy after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Average of one key accuracy indicator from each of 9 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, psychomotor vigilance)
Morning neurobehavioural accuracy after exposure to pink noise | In the morning immediately after the Pink noise night
  Average of one key accuracy indicator from each of 9 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, psychomotor vigilance)
Morning neurobehavioural accuracy after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Average of one key accuracy indicator from each of 9 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, psychomotor vigilance)
Baseline evening neurobehavioural speed | In the evening of the day following the Control night
  Average of one key speed indicator from each of 10 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance)
Evening neurobehavioural speed after exposure to nocturnal traffic | In the evening of the day following the Traffic noise night
  Average of one key speed indicator from each of 10 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance)
Evening neurobehavioural speed after exposure to pink noise | In the evening of the day following the Pink noise night
  Average of one key speed indicator from each of 10 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance)
Evening neurobehavioural speed after exposure to nocturnal traffic and pink noise | In the evening of the day following the Traffic noise + pink noise night
  Average of one key speed indicator from each of 10 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance)
Baseline evening neurobehavioural accuracy | In the evening of the day following the Control night
  Average of one key speed indicator from each of 9 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, psychomotor vigilance)
Evening neurobehavioural accuracy after exposure to nocturnal traffic | In the evening of the day following the Traffic noise night
  Average of one key speed indicator from each of 9 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, psychomotor vigilance)
Evening neurobehavioural accuracy after exposure to pink noise | In the evening of the day following the Pink noise night
  Average of one key speed indicator from each of 9 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, psychomotor vigilance)
Evening neurobehavioural accuracy after exposure to nocturnal traffic and pink noise | In the evening of the day following the Traffic noise + pink noise night
  Average of one key speed indicator from each of 9 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, psychomotor vigilance)
Baseline Ethanol concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Trimethylamine-N-oxide concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline 2-Aminobutyric acid concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Alanine concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Asparagine concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Creatine concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Creatinine concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Glutamic acid concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Glutamine concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Glycine concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Histidine concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Isoleucine concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Leucine concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Lysine concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Methionine concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline N,N-Dimethylglycine concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Ornithine concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Phenylalanine concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Proline concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Sarcosine concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Threonine concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Tyrosine concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Valine concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline 2-Hydroxybutyric acid concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Acetic acid concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Citric acid concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Formic acid concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Lactic acid concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Succinic acid concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Choline concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline 2-Oxoglutaric acid concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline 3-Hydroxybutyric acid concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Acetoacetic acid concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Acetone concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Pyruvic acid concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline D-Galactose concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Glucose concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Glycerol concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Baseline Dimethylsulfone concentration (mmol/L) | In the morning immediately after the Control night
  Determined from NMR analysis of blood plasma
Ethanol concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Trimethylamine-N-oxide concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
2-Aminobutyric acid concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Alanine concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Asparagine concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Creatine concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Creatinine concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Glutamic acid concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Glutamine concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Glycine concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Histidine concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Isoleucine concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Leucine concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Lysine concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Methionine concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
N,N-Dimethylglycine concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Ornithine concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Phenylalanine concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Proline concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Sarcosine concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Threonine concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Tyrosine concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Valine concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
2-Hydroxybutyric acid concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Acetic acid concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Citric acid concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Formic acid concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Lactic acid concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Succinic acid concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Choline concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
2-Oxoglutaric acid concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
3-Hydroxybutyric acid concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Acetoacetic acid concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Acetone concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Pyruvic acid concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
D-Galactose concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Glucose concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Glycerol concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Dimethylsulfone concentration (mmol/L) after exposure to nocturnal traffic | In the morning immediately after the Traffic noise night
  Determined from NMR analysis of blood plasma
Ethanol concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Trimethylamine-N-oxide concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
2-Aminobutyric acid concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Alanine concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Asparagine concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Creatine concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Creatinine concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Glutamic acid concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Glutamine concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Glycine concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Histidine concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Isoleucine concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Leucine concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Lysine concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Methionine concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
N,N-Dimethylglycine concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Ornithine concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Phenylalanine concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Proline concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Sarcosine concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Threonine concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Tyrosine concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Valine concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
2-Hydroxybutyric acid concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Acetic acid concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Citric acid concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Formic acid concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Lactic acid concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Succinic acid concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Choline concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
2-Oxoglutaric acid concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
3-Hydroxybutyric acid concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Acetoacetic acid concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Acetone concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Pyruvic acid concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
D-Galactose concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Glucose concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Glycerol concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Dimethylsulfone concentration (mmol/L) after exposure to nocturnal pink noise | In the morning immediately after the Pink noise night
  Determined from NMR analysis of blood plasma
Ethanol concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Trimethylamine-N-oxide concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
2-Aminobutyric acid concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Alanine concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Asparagine concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Creatine concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Creatinine concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Glutamic acid concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Glutamine concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Glycine concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Histidine concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Isoleucine concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Leucine concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Lysine concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Methionine concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
N,N-Dimethylglycine concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Ornithine concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Phenylalanine concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Proline concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Sarcosine concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Threonine concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Tyrosine concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Valine concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
2-Hydroxybutyric acid concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Acetic acid concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Citric acid concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Formic acid concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Lactic acid concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Succinic acid concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Choline concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
2-Oxoglutaric acid concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
3-Hydroxybutyric acid concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Acetoacetic acid concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Acetone concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Pyruvic acid concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
D-Galactose concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Glucose concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Glycerol concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma
Dimethylsulfone concentration (mmol/L) after exposure to nocturnal traffic and pink noise | In the morning immediately after the Traffic noise + pink noise night
  Determined from NMR analysis of blood plasma

SECONDARY OUTCOMES:
Cardiovascular activation in response to noise | Event-related, occurring within the time window of each discrete noise event, during each of the five study nights (23:00 to 07:00)
  Change in heart rate (ECG)
Evening subjective sleepiness, assessed using the Karolinska Sleepiness Scale | Every study evening
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Morning subjective sleepiness, assessed using the Karolinska Sleepiness Scale | Every study morning
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Evening auditory fatigue | Every study evening
  Perceived auditory fatigue, self-reported on a 5-point verbal scale, from 1 - "Not at all" (best outcome) to 5 - "Extremely" (worst outcome)
Morning auditory fatigue | Every study morning
  Perceived auditory fatigue, self-reported on a 5-point verbal scale, from 1 - "Not at all" (best outcome) to 5 - "Extremely" (worst outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Smith, PhD, Principal Investigator — Göteborg University
Locations (1):
- University of Gothenburg, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vincens N, Nause A, Basner M, Fredriksson S, Malmodin D, Bay Nord A, Persson Waye K, Younes M, Zou D, Smith MG. Pink noise reduces impact of traffic noise on sleep and the blood metabolome: a cross-over pilot study. Commun Med (Lond). 2026 Jan 10. doi: 10.1038/s43856-026-01380-5. Online ahead of print. PMID 41513961